CLINICAL TRIAL: NCT02726503
Title: Phase II Study Assessing the Efficacy and Safety of Lenvatinib for Anaplastic Thyroid Cancer (HOPE)
Brief Title: Phase II Study Assessing the Efficacy and Safety of Lenvatinib for Anaplastic Thyroid Cancer
Acronym: HOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRIHN1504; UMIN000020773 (Other: UMIN-CTR)
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: anaplastic thyroid cancer, lenvatinib
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — All patients will receive lenvatinib 24 mg orally once daily at almost the same time. The treatment will be started within 1 week after enrollment. 1 cycle consists of 4 weeks.
  The administration will be continued until patients meet withdrawal criteria. If any toxicity manifested that cannot be ruled out causal association with the study drug, drug withdrawal or dosage reduction will be conducted in accordance with drug withdrawal/dosage reduction criteria.

SUMMARY:
The purpose of this phase Ⅱ study is to assess the efficacy and safety of lenvatinib for anaplastic thyroid cancer patients who are diagnosed as unresectable. The total duration of the study will be 30 months. All patients will start administration of lenvatinib within 1 week of enrollment and receive the study drug 24mg orally once daily at almost the same time. 1 cycle consists of 4 weeks. Treatment term starts on the day 1st of drug administration of cycle 1 and administration will be continued until patients meet withdrawal criteria. Safety and efficacy assesment will be conducted on a regular basis during the trial. Tumor evaluation will be conducted at 4weeks, 8 weeks, 12 weeks, 16 weeks and at every 8 weeks after the 16th week since initial administration. When study drug administration terminated,tests of the drug termination will be conducted within 7 days of withdrawal and final observation will be conducted at 30 days after the last dose. Survival survey will be conducted at follow-up term. After the termination of the study drug, survival follow up survey will be conducted every 12 weeks unless patients withdraw enrollment of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed as anaplastic thyroid cancer
2. Unresectable disease
3. Have measurable lesion defined by the RECIST version 1.1
4. Have adequate organ function and meet following laboratory value:

   1. Bone marrow function test within 14 days prior to enrollment:

      neutrophil count>=1.5 x 103/microL blood platelet count>=10.0 x 104/microL hemoglobin amount>=9.0 g/dL
   2. Liver function test within 14 days prior to enrollment:

      AST,ALT<=3.0 x ULN(without liver metastatic) AST,ALT<=5.0 x ULN(with liver metastatic) bilirubin<=2.0 mg/dL
   3. Kidney function test within 14 days prior to enrollment:

      GFR estimation>=50 ml/min/1.73 m2 GFR estimation calculated by following formula. Male:194 x(serum creatinine concentration)-1.094 x(Age)-0.287 Female:Male GFR estimation x 0.739
   4. Cardiac function test within 28 days prior to enrollment: 12-lead electrocardiogram: no clinically important abnormality as shown below: heart disease, severe arrhythmia etc.
5. Regardless of usage of antihypertensive drug, systolic blood pressure <=140 mm Hg and diastolic blood pressure <=90 mm Hg (If already taking antihypertensive drug, must have capacity of further antihypertensive therapy.)
6. ECOG performance status 0-2
7. Ability to swallow oral medications
8. Life expectancy greater than 8 weeks
9. Have signed written informed consent to participate in this study

Exclusion Criteria:

1. Have complications or medical history of

   1. Complication of brain metastasis (Exclude if cured and in clinically stable condition for more than 1 month prior to screening.)
   2. Treatment required complication of systemic infectious disease
   3. Complication of pulmonary fibrosis or interstitial pneumonitis
   4. Medical history of clinically significant cardiovascular disease within 6 months of initial dose as: NYHA class above 2 leveled congestive heart failure, unstable angina, cardiac infarction or cardiac arrhythmia with paroxysmal or required treatment e) Uncontrollable complication of diabetes mellitus f) hemoptysis within 3 weeks of enrollment (blood volume of more than half of teaspoon) g) Medical history of hemorrhagic or thrombotic disease within 6 months of enrollment h) If proteinuria values above 2+ by urinary protein qualitative test, conduct 24-hour urine collection and the urine protein determined as 1g/24 hours or more. (can substitute to the ratio of proteinuria in morning urine/creatinine) i) Malabsorption at gastrointestinal tract and any of the complication diseases that investigator considers that will be affected to lenvatinib absorption j) Recent major surgery within 2 weeks (if needle biopsy within 1 week) of enrollment k) Drainage required celomic fluid stagnation
2. Have history of lenvatinib administration
3. Confirmed tumor invasion to the carotid arteries
4. Have history of high dose external radiation therapy to cervical region, and irradiated tumor location close to the carotid arteries.
5. Have any unresolved toxicity greater than 1 by CTCAE v4.0.
6. Have active double cancer
7. Female patients who are pregnant, lactating, breast feeding or have childbearing potential
8. Psychiatric disorder and regarded by the investigator as inadequate for this study enrollment
9. Confirmed as no resistance to any component of this drug
10. Currently receiving other interventional clinical study treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2016-04-04 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 30 months
  OS is defined as time frame from date of initial dose until date of death from any cause. Or until the last confirmed survival date, study cut-off date which ever comes first.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to 30 months
  PFS is defined as time frame from date of initial dose until the date of first confirmed disease progression, until date of death from any cause or the last tumor evaluating date whichever comes first.
Best Overall Response (BOR) | up to 30 months
  BOR is defined as the best total efficacy record during the date of initial dose to the date of study completion, by which evaluated with following index. Complete Response (CR), Partial Response (PR), Stable Disease (SD is defined as ≧3 weeks),Pharmacodynamics/Progressive Disease (PD) or Not Evaluable (NE).
Objective Response Rate (ORR) | up to 30 months
  ORR is defined as the ratio of patients who are evaluated as CR or PR in Best Overall Response (BOR).
Disease Control Rate (DCR) | up to 30 months
  DCR is defined as the ratio of patients who are evaluated as CR, PR or SD in Best Overall Response (BOR).
Clinical Benefit Rate (CBR) | up to 30 months
  CBR is defined as the ratio of patients who are evaluated as CR, PR or durable SD (dSD is defined as ≧11 weeks SD) in Best Overall Response (BOR).
Safety assessment on the incidence ratio of adverse events | up to 30 months
  Safety assessment will be assessed by the ratio of adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Iwao Sugitani, M.D., Ph.D, Study Director — Graduate School of Medicine Nippon Medical School; Makoto Tahara, M.D., Ph.D, Study Director — National Cancer Center Hospital East
Locations (23):
- Japan (23):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - IUHW Ichikawa Hospital, Ichikawa, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Japanese Red Cross Narita Hospital, Narita, Chiba
  - Kuma Hospital, Kobe, Hyōgo
  - Kobe Univbersity Hospital, Kobe, Hyōgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Miyaghi Cancer Center, Natori-shi, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinsyu University School of Medicine Department of Surgery, Matsumoto, Nagano
  - Nara Hospital Kinki University Faculty of Medicine, Ikoma, Nara
  - Nara Medical University, Kashihara, Nara
  - Osaka Police Hospital, Osaka, Osaka
  - Osaka City University Graduate School of Medicine and Faculty of Medicine, Osaka, Osaka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Ito Hospital, Shibuya-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo